CLINICAL TRIAL: NCT04877847
Title: Low Frequency Therapeutic Ultrasound System Pivotal Clinical Trial
Brief Title: Multi-Center Trial Utilizing Low Frequency Ultrasound in the Prevention of Post-Contrast Acute Kidney Injury
Acronym: LOTUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Sonogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP-001
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Contrast-induced Nephropathy; Chronic Kidney Diseases
Keywords: coronary arteriography; nitric oxide
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: A total of up to 234 participants will be randomized 2:1
Who Masked: Participant, Care Provider
Masking Description: Participant and clinical staff will be blinded to which arm the participant is randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Low-Frequency Therapeutic Ultrasound (Experimental): LOTUS system will be operated per operated per normal instructions
  Interventions: Device: Low-frequency therapeutic ultrasound (LOTUS)
- Sham Control (Sham Comparator): LOTUS system will be set to Control setting
  Interventions: Device: LOTUS System with Ultrasound Disabled

INTERVENTIONS:
Device: Low-frequency therapeutic ultrasound (LOTUS) — Participants will wear low-frequency therapeutic ultrasound system for procedure. Device will be turned on per normal operating instructions.
  Arms: Low-Frequency Therapeutic Ultrasound
Device: LOTUS System with Ultrasound Disabled — Participants will wear low-frequency therapeutic ultrasound system for procedure. Device will be turned on and set to Control Setting.
  Arms: Sham Control

SUMMARY:
Multi-center randomized trial to assess the safety and performance of low-frequency therapeutic ultrasound for maintaining renal function after contrast exposure.

DETAILED DESCRIPTION:
This is a multi-center, randomized, controlled clinical trial designed to assess the safety and performance of the Sonogenix RENOBOOST as an adjunctive therapy for maintaining renal function after contrast exposure. The trial will enroll up to 234 subjects not taking oral nitrates and at high-risk of developing PC-AKI undergoing coronary arteriography for a planned percutaneous coronary intervention in up to 10 clinical sites in the US and up to 3 clinical sites outside the US.

All subjects will be pre- treated with 0.9 percent NaCl at 3 ml/kg/h 1 hour before and 1 ml/kg/h during and 6 hours post procedure. Participants will be randomized in a 2:1 fashion to either active adjunctive therapy with the Sonogenix RENOBOOST or sham control.

Subjects will have clinical follow-up examination 30 days post index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant is greater than or equal to 18 years
* Baseline renal dysfunction defined as one of the following:

  1. eGFR greater than 30
  2. eGFR 30-45, with or without risk factors for AKI defined as diabetes mellitus, congestive heart failure, proteinuria (defined as albuminuria greater than 300mg/day).
  3. eGFR 45-60, with at least one risk factor for AKI defined as diabetes mellitus, congestive heart failure, proteinuria (defined as albuminuria greater than 300mg/day).
* Participant is presenting for a planned percutaneous coronary intervention (PCI)
* Participant scheduled to undergo cardiac catheterization including coronary arteriography that is anticipated to require at least 100 ml of iso-osmolar or low- osmolar contrast, and that is anticipated to include single-vessel stent implantation that does not include chronic total occlusion.
* Participant had not been hospitalized or treated for a change in renal function within 30 days of enrollment.
* Participant has provided written informed consent.
* Participant is willing to comply with study follow-up requirements.

Exclusion Criteria

* Participant is anuric or currently undergoing renal replacement therapy.
* Participant is currently taking oral nitrates.
* Participant is undergoing a procedure requiring selective cannulation and injection of contrast into the renal arteries.
* Participant presented with ST-segment elevation myocardial infarction.
* Participant has a metal implant in the hip or lumbar spine.
* Participant received or is anticipated to receive additional intravenous or intraarterial contrast from 7 days prior to cardiac catheterization to 4 days after cardiac catheterization.
* Addition, discontinuation, or dose change of angiotensin-converting enzyme inhibitor, angiotensin receptor blocker, diuretic, trimethoprim, non-steroidal anti-inflammatory drugs, cimetidine, or metoclopramide with 7 days prior to cardiac catheterization.
* Participant has a known allergy to contrast medium that cannot be adequately pre-medicated.
* Participant has new-onset heart failure with New York Heart Association (NYHA) classification of III or IV within 30 days prior to the index procedure.
* Recent stroke within 90 days prior to the index procedure.
* Participant has known or suspected active infection at the time of the index procedure.
* Participant is pregnant and/or breast-feeding or intends to become pregnant during the time of the study.
* Participant is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol.
* Participant is known to be incarcerated, mentally incompetent, and/or alcohol or drug abuser.
* Participant is participating in another investigational drug or medical device study that has not completed primary endpoint(s) evaluation or clinically interferes with the endpoints from this study or subject is planning to participate in such studies prior to the completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 48 hours
  Incidence of acute kidney injury (AKI) defined as a greater than 0.3 mg/dl increase in serum creatinine (SCr)
Primary Safety Endpoint | 30 days
  Composite of all Adverse Events (AE) including RENOBOOST (device) related adverse events, and major adverse events (MAE)

SECONDARY OUTCOMES:
Incidence of Post Contrast Acute Kidney Injury | at 72 hours post-contrast exposure or need for renal replacement therapy (RRT)
  defined as greater than or equal to 0.3 mg/dl or greater than or equal to 25 percent rise in SCr
Incidence of Post Contrast Acute Kidney Injury | at 72 hours post-contrast exposure or need for renal replacement therapy (RRT)
  defined as greater than or equal to 0.5 mg/dl or greater than or equal to 25 percent rise in SCr
Incidence of contrast-induced nephropathy | within 96 hours post-contrast exposure or need for RRT
  defined as greater than or equal to 0.3 mg/dl or greater than or equal to 25 percent rise in SCr
Occurrence of (stage 1, 2, or 3) acute kidney injury (AKI) | within 30 days after index procedure
  defined as greater than or equal to 2-fold rise in SCr, increase in SCr to greater than or equal to 4.0 mg/dl, or initiation of RRT
Incidence of Post Contrast Acute Kidney Injury | within 96 hours post-contrast exposure or need for RRT
  defined as greater than or equal to 0.3 mg/dl or greater than or equal to 25 percent rise in SCr
Occurrence of (stage 1, 2, or 3) acute kidney injury (AKI) | within 96 hours of index procedure
  defined as Stage 1 - Serum Creatinine 1.5-1.9 times baseline or greater than or equal to 0.3 mg/dL increase, Stage 2 - Serum Creatinine 2-2.9 times baseline, Stage 3 - Serum Creatinine 3 times baseline or Increase in serum creatinine to greater than or equal to 4 mg/dL or Initiation of renal replacement therapy
Maximum percent-change | within 96 hours after contrast exposure
  Maximum percent-change in SCr
Absolute and percent-change in estimated glomerular filtration rate (eGFR) | from baseline within 96 hours after contrast exposure.
  as calculated using the Modification of Diet in Renal Disease Study Group (MDRD)
Total urine output | through baseline procedure
  defined as the amount of urine collected in cc/hour.
Hospitalization | following the baseline procedure through discharge from the hospital up to 30 days
  Hospital length of stay
Intensive Care | following the baseline procedure through discharge from the Intensive Care Unit up to 30 days
  Intensive care unit length of stay

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Henry Ford Hopsital, Detroit, Michigan
  - McLaren Northern Michigan, Petoskey, Michigan
  - University of Pennsylvania Medical Center, Pittsburgh, Pennsylvania
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No